CLINICAL TRIAL: NCT05646056
Title: A Noninterventional, Single-Center Feasibility Study to Evaluate Longitudinal Measures of Heart Failure Risk Using the Pyxida System
Brief Title: A Noninterventional, Single-Center Feasibility Study to Evaluate Measures of Heart Failure Risk
Status: Completed | Type: Observational
Sponsor: Prolaio (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-001-001
Record Dates: First submitted 2022-11-23; First posted 2022-12-12 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Cardiomyopathy, Hypertrophic; Left Ventricular Hypertrophy
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Healthy subjects
  Interventions: Device: Software
- Asymptomatic subjects with a history of left ventricular hypertrophy (LVH) and NYHA Class I
  Interventions: Device: Software
- Asymptomatic subjects with a history of heart failure (HF) and NYHA Class I
  Interventions: Device: Software
- Subjects with a history of hypertrophic cardiomyopathy (HCM) and NYHA Class I, II
  Interventions: Device: Software

INTERVENTIONS:
Device: Software — Observation only

SUMMARY:
This is a non-invasive/observational study in healthy and mild HF subjects utilizing clinical and ambulatory measurements to improve detection, monitoring, and management of HF risks.

ELIGIBILITY:
Key Inclusion Criteria:

* Cohort 2: Confirmed medical history of LVH based on American College of Cardiology (ACC)/American Heart Association (AHA) guidelines and NYHA Class I at screening
* Cohort 3: Confirmed medical history of HF consistent with current ACC/AHA guidelines and NYHA Class I at screening
* Cohort 4: Confirmed medical history of HCM consistent with ACC/AHA guidelines and NYHA Class I or II at screening

Key Exclusion Criteria:

* Active neurological disorder, such as uncontrolled seizure disorder.
* Current diagnosis of cancer or other known acute chronic infection, such as hepatitis B or hepatitis C, by medical history or an active infection requiring interventional therapy at screening.
* Shortness of breath, fatigue, heart palpitations, pain, or other limitations of physical activity

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Single-center study of asymptomatic healthy subjects and subjects with HF risk factors and no more than mild to moderate symptoms
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of the Pyxida System to collect measurements of heart failure (HF) risk | 14 days
  Percentage of complete daily datasets transmitted to the Pyxida System database at the end of the monitoring period

SECONDARY OUTCOMES:
To evaluate subject compliance and experience using the Pyxida System | 14 days
  Outcomes of subject post-study survey

OTHER OUTCOMES:
To evaluate the relationship between in-clinic and ambulatory measures using the Pyxida System | 14 days
  Correlation between in-clinic 6-minute walk test (6MWT) measures of exercise tolerance and ambulatory electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koren, MD, Principal Investigator — Jacksonville Center For Clinical Research
Locations (1):
- Jacksonville Center for Clinical Research, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided